CLINICAL TRIAL: NCT00771251
Title: A Study of Golimumab (CNTO148) Monotherapy in Patients With Active Rheumatoid Arthritis
Brief Title: A Safety and Efficacy Study of Golimumab (CNTO148) in Patients With Active Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR015343; JNS012-JPN-04 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Fully Human anti-TNFa monoclonal antibody; CNTO148; Golimumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CNTO 148 50 mg (Experimental)
  Interventions: Drug: CNTO 148
- CNTO 148 100 mg (Experimental)
  Interventions: Drug: CNTO 148
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNTO 148 — 50 mg or 100 mg given as a subcutaneous (under the skin) injection once every 4 weeks up to Week 116.
  Other Names: Golimumab
  Arms: CNTO 148 100 mg; CNTO 148 50 mg
Drug: Placebo — Placebo identical in appearance to CNTO 148 given as a subcutaneous (under the skin) injection once every 4 weeks until week 12 and then CNTO148 50mg SC injections every 4 weeks from week 16 until week 116.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of golimumab in patients with active rheumatoid arthritis despite DMARD (Disease-modifying antirheumatic drugs) therapy. Another objective is to evaluate the pharmacokinetics of golimumab.

DETAILED DESCRIPTION:
This study is designed as a placebo-controlled study of golimumab monotherapy for the purpose of demonstrating the safety and effectiveness of golimumab, a new, fully human anti-TNF (Tumor necrosis factor) a monoclonal antibody produced by mean of HuMab mouse technology. Other reasons for using the study design are as follows: the effects of golimumab given alone must be confirmed as in the case of other drugs; and golimumab may be used even in patients not on the treatment with methotrexate (MTX). There will be 3 treatment groups in the study as follows: CNTO148 50 mg group, CNTO 148 100 mg group, and Placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with rheumatoid arthritis at least 3 months prior to registration and who are definitely identified as having rheumatoid arthritis, at the time of informed consent, according to the criteria for classification established by the American College of Rheumatology (1987)
* Patients who have previously not responded to at least one DMARD (before informed consent is obtained)
* Patients who, if they are on the treatment with a DMARD, the DMARD can be washed out for at least 4 weeks before the first administration
* Patients having at least 6 swollen joints and 6 tender joints at the time of registration and immediately before the first injection

Exclusion Criteria:

* Patients with a history of hypersensitivity to human immunoglobulin proteins or other ingredients of golimumab
* Patients who have previously experienced or are suffering from any of the following diseases: (i) Collagen diseases other than rheumatoid arthritis, (ii) Latent or active granulomatous infections such as histoplasmosis and coccidioidomycosis, (iii) Felty syndrome, etc
* Patients with a severe, advanced, or poorly controlled disease in any of the kidney, liver, blood, gastrointestinal system, endocrine system, lung, heart, nervous system, psychiatric system, and brain

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2008-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
ACR 20% response | Weel 14

SECONDARY OUTCOMES:
ACR 50% response, ACR 70% response, ACR 90% response, Changes from the pretreatment values in the DAS (Disease Activity Score) 28, and the HAQ (Health assessment questionnaire) | Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (67):
- Japan (67):
  - Asahikawa
  - Ayauta
  - Azumino
  - Chiba
  - Fuchū
  - Fukui
  - Fukuoka
  - Fukushima
  - Gifu
  - Goshogawara
  - Hachiōji
  - Hamamatsu
  - Higashi-Hiroshima
  - Hiki
  - Hiroshima
  - Hitachi
  - Hitachi-Naka
  - Iruma
  - Izumisano
  - Izumo
  - Kamakura
  - Katō
  - Kawachi-Nagano
  - Kawagoe
  - Kawasaki
  - Kita-Gun
  - Kitakyushu
  - Kitamoto
  - Kobe
  - Kumamoto
  - Kyoto
  - Matsue
  - Matsumoto
  - Matsuyama
  - Nagano
  - Nagoya
  - Narashino
  - Niigata
  - Nishinomiya
  - Ohta-Ku
  - Osaka
  - Ōita
  - Ōsaka-sayama
  - Ōsaki
  - Sagamihara
  - Saitama
  - Sapporo
  - Sasebo
  - Sendai
  - Shimotsuga
  - Shimotsuke
  - Shinjuku-Ku
  - Shizuoka
  - Suita
  - Tokushima
  - Tokyo
  - Tomigusuku
  - Toshima-Ku
  - Toyama
  - Toyoake
  - Toyohashi
  - Tsu
  - Tsukuba
  - Tsukubo
  - Ube
  - Yokohama
  - Yufu

REFERENCES:
- [Result] Takeuchi T, Harigai M, Tanaka Y, Yamanaka H, Ishiguro N, Yamamoto K, Miyasaka N, Koike T, Kanazawa M, Oba T, Yoshinari T, Baker D; GO-MONO study group. Golimumab monotherapy in Japanese patients with active rheumatoid arthritis despite prior treatment with disease-modifying antirheumatic drugs: results of the phase 2/3, multicentre, randomised, double-blind, placebo-controlled GO-MONO study through 24 weeks. Ann Rheum Dis. 2013 Sep 1;72(9):1488-95. doi: 10.1136/annrheumdis-2012-201796. Epub 2012 Sep 14. PMID 22984173
- See also: A Study of Golimumab (CNTO148) monotherapy in Patients with Active Rheumatoid Arthritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=427&filename=CR015343_CSR.pdf